CLINICAL TRIAL: NCT01931228
Title: Contribution of Mechanical Insufflation-Exsufflation in Preventing Respiratory Failure Post Extubation in Patient With Critical Care Neuromyopathy
Brief Title: Mechanical Insufflation-Exsufflation in Preventing Post Extubation Respiratory Failure in Patient With Critical Care Neuromyopathy
Acronym: NEUROMIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUBX 2011/21
Record Dates: First submitted 2013-08-22; First posted 2013-08-29 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Acute Respiratory Insufficiency; Respiratory Failure
Keywords: Intensive care unit; acute respiratory insufficiency; Respiratory failure; Mechanical Insufflation-Exsufflation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MI-E plus manually assisted coughing (Experimental)
  Interventions: Procedure: MI-E plus manually assisted coughing
- Manually assisted coughing only (Experimental)
  Interventions: Procedure: manually assisted coughing

INTERVENTIONS:
Procedure: MI-E plus manually assisted coughing — MI-E plus manually assisted coughing twice a day for 48h after extubation. After this period and before discharge of the icu or day28 maximum, patients received only one daily session.
  Arms: MI-E plus manually assisted coughing
Procedure: manually assisted coughing — Manually assisted coughing twice a day for 48h after extubation. After this period and before discharge of the icu or day28 maximum, patients received only one daily session.
  Arms: Manually assisted coughing only

SUMMARY:
Respiratory failure after extubation is a relevant consequence of poor airway clearance due to respiratory muscle weakness and respiratory failure after extubation and reintubation is associated with increased morbidity and mortality.

the study will evaluate the contribution of Mechanical Insufflation-Exsufflation (MI-E) in Preventing Respiratory Failure After Extubation as compared manually assisted coughing

DETAILED DESCRIPTION:
Critical Care Neuromyopathy (CCN) occur in 25% of patient in Intensive Care Unit (ICU). Respiratory failure after extubation is a relevant consequences of poor airway clearance due to respiratory muscle weakness. Respiratory failure is a major cause for reintubation which increase severity of illness, this is an independent risk factor for nosocomial pneumonia, increased hospital stay and mortality. Currently, respiratory physiotherapy includes, manual expiration assist often associated with nasotracheal aspiration. Despite of this care, respiratory failure occur in 30% of patients within 48 after planned extubation. MI-E has been evaluated for neuromuscular disease patient, and increase peak cough flow and the airway clearance. So the beneficials effects of MI-E should be confirmed in a trial in this specific population.

We planned to conduct a study evaluating the efficacy of MI-E in the prevention of extubation failure and mortality in these patients. If no signs of respiratory failure appeared after 120 min of a spontaneous breathing trial, patients will be extubated and randomly allocated after extubation to MI-E group or control group. The clinical follow-up will be as follow: the incidence of extubation failure, the reintubation, the ICU or 28-day survival,90-day survival, ICU length of stay.

ELIGIBILITY:
Inclusion criteria:

* Male or female patient aged ≥ 18 years.
* Patient admitted in participant ICU.
* Patient intubated for 48 hours at least.
* Patient presenting an ICU acquired neuromuscular disorders.

Exclusion criteria:

* Respiratory or haemodynamic instability.
* Patient having a contraindication to use face mask (Recent facial surgery, severe craniofacial trauma,…) gastroesophageal surgery.
* Severe ventricular rhythm disorders.
* Patient with tracheotomy.
* Uncontrollable vomiting.
* Severe sepsis.
* Upper airway disorders.
* Upper gastrointestinal bleeding.
* Any decision to limit therapeutic effort in the ICU.
* Patient with limit therapeutic effort in the ICU with unsuccessful spontaneous respiratory trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2012-05-03 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Incidence of respiratory failure after extubation | 48h post extubation (48h after inclusion)

SECONDARY OUTCOMES:
the increase in peak cough flow | End of intensive care or day 28 after inclusion
the incidence of reintubation | End of intensive care or day 28 after inclusion
the average time of hospitalization in the intensive care unit | End of intensive care or day 28 after inclusion
the incidence of nasotracheal suction | End of intensive care or day 28 after inclusion
the number of additional physiotherapy sessions | End of intensive care or day 28 after inclusion
the ICU mortality or 28-day survival | 28 days after inclusion
90 days survival | 90 days after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Philippe WIBART, Physical therapist, Principal Investigator — University Hospital, Bordeaux; Antoine BENARD, MD, Study Chair — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France

REFERENCES:
- [Derived] Wibart P, Reginault T, Garcia-Fontan M, Barbrel B, Bader C, Benard A, Parreira VF, Gonzalez-Anton D, Bui NH, Gruson D, Hilbert G, Martinez-Alejos R, Vargas F. Effects of mechanical in-exsufflation in preventing postextubation acute respiratory failure in intensive care acquired weakness patients: a randomized controlled trial. Crit Care Sci. 2023 Apr-Jun;35(2):168-176. doi: 10.5935/2965-2774.20230410-en. PMID 37712806